CLINICAL TRIAL: NCT04834414
Title: CHIlled Platelet Study
Brief Title: CHIlled Platelet Study "CHIPS"
Acronym: CHIPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philip Spinella (Other)
Collaborators: University of Utah (Other); University of Minnesota (Other); Washington University School of Medicine (Other); United States Department of Defense (U.S. Federal Agency); University of Pittsburgh (Other)
Responsible Party: Sponsor-Investigator, Philip Spinella, Professor- Surgery and Critical Care Medicine, Co- Director- Trauma and Transfusion Medicine Research Center, Associate Medical Director- Center for Military Medicine Research, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CHIPS; W81XWH2090021 (Other Grant/Funding Number: DoD)
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Blood Loss
Keywords: platelets; cold-stored platelets; bleeding; hemostasis; complex cardiac surgery
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Adaptive Design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Partial Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Room Temperature Platelets (Active Comparator): Platelets stored at 20-24 degrees Celsius
  Interventions: Biological: Room Temperature Platelets
- Cold Stored Platelets (Experimental): Platelets stored at 1-6 degree Celsius
  Interventions: Biological: Cold Stored Platelets

INTERVENTIONS:
Biological: Cold Stored Platelets — Platelets stored at 1-6 degree Celsius
  Arms: Cold Stored Platelets
Biological: Room Temperature Platelets — Platelets stored at 20-24 degrees Celsius
  Arms: Room Temperature Platelets

SUMMARY:
A phase 3 randomized partial blind storage duration ranging study in patients undergoing complex cardiac surgery that will compare the transfusion of cold stored platelets to standard room temperature stored platelets. The primary objective is to establish that cold stored platelets have a non-inferiority (or superiority) to room temperature platelets.

ELIGIBILITY:
Inclusion Criteria:

* Viable neonates ≥ 3 kg at time of enrollment (as defined in Section 4.1) OR age greater than 28 days and less than 85 years of age at time of consent; AND
* Planned complex cardiac surgery with planned use of cardiopulmonary bypass, with an expectation of bleeding requiring platelet transfusion.

Exclusion Criteria:

* Expected order for washed or volume reduced platelets
* Patient with known anti-platelet antibodies
* Platelet transfusion refractoriness due to anti-HLA antibodies
* Known or suspected pregnancy
* Previously randomized in this study
* Conscious objection or unwillingness to receive blood products
* Known IgA deficiency
* Known congenital platelet disorder
* Known congenital bleeding disorder
* Planned post-operative extracorporeal membrane oxygenation (ECMO), ventricular assist device (VAD), and/or continuous renal replacement therapy (CRRT)/ hemodialysis
* Patients intended to receive whole blood either intra-operative or post-operative for bleeding
* Platelet transfusion (of any type) within 24 hours prior to the date of surgery
* Pre-operative thrombocytopenia, defined as platelet count <75x10(9)/L, based on the most recent labs completed within 72 hours prior to the date of surgery.

Ages: 0 Days to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Hemostatic efficacy | 24 hours after first study platelet transfusion
  Assessed by a bleeding score, a modified Peri-Operative bleeding score: the score ranges from 1-5. A lower score signifies a better outcome.

SECONDARY OUTCOMES:
Chest tube output | 24 hours from first study platelet transfusion or ICU admit (determined from which occurs last)
  Assessed by volume

OTHER OUTCOMES:
Blood product administration | 24 and 72 hours from start time of first study platelet transfusion
  The quantity of RBCs, Plasma, Platelets, Cryoprecipitate, and Whole blood
Total Dose of individual hemostatic adjuncts | 24 and 72 hours from start time of first study platelet transfusion
  Antifibrinolytic and coagulation factor concentrates
Mechanical ventilation | up to 28 days after first study platelet transfusion
  Duration of mechanical ventilation days
Length of stay | up to 28 days
  ICU and hospital length of stay
Relative change in hemostatic parameters | 6 and 24 hours after first study platelet transfusion
  CBC (platelet count and hemoglobin), PT/INR, PTT, fibrinogen, and TEG
Unplanned sternal closure delay | prior to ICU admission
  Sternum left open after cardiac surgery
Re-exploration for bleeding | 24 hours first study platelet transfusion
  Return to OR after ICU admission
Unplanned extracorporeal support post operatively | within 48 hours of first study platelet transfusion
  Placed on ECMO
Morbidities after ICU admission | within 7 days of first study platelet transfusion
  Acute respiratory distress syndrome, need for and duration of renal support, renal failure, septic shock
Measures of end organ injury | within 48 hours of first study platelet transfusion
  If BUN, creatinine, lactate, troponin, alanine aminotransferase (ALT) are collected clinically.
Transfusion associated adverse events | within 7 days of first study platelet transfusion
  As per CDC guidelines
Arterial thrombotic event | within 7 days of first study platelet transfusion
  Stroke, MI
Venous thrombotic event | within 7 days of first study platelet transfusion
  Deep vein thrombosis or pulmonary embolism confirmed by ultrasound, venography, perfusion scan, spiral CT, MRI, or pulmonary angiogram
All cause mortality | up to 28 days
  Death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Philip C Spinella, MD, Study Director — University of Pittsburgh; Marie E Steiner, MD, Study Director — University of Minnesota; Nicole D Zantek, MD, Study Director — University of Minnesota
Locations (27):
- United States (25):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola Universtiy Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - John Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Children's Medical Center, Dallas, Texas
  - University of Texas Medical Center Clements, Dallas, Texas
  - Baylor Texas Children's, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Wisconsin- Madison, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Australia (2):
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krachey E, Viele K, Spinella PC, Steiner ME, Zantek ND, Lewis RJ. The design of an adaptive clinical trial to evaluate the efficacy of platelets stored at low temperature in surgical patients. J Trauma Acute Care Surg. 2018 Jun;84(6S Suppl 1):S41-S46. doi: 10.1097/TA.0000000000001876. PMID 29521797
- [Background] Strandenes G, Sivertsen J, Bjerkvig CK, Fosse TK, Cap AP, Del Junco DJ, Kristoffersen EK, Haaverstad R, Kvalheim V, Braathen H, Lunde THF, Hervig T, Hufthammer KO, Spinella PC, Apelseth TO. A Pilot Trial of Platelets Stored Cold versus at Room Temperature for Complex Cardiothoracic Surgery. Anesthesiology. 2020 Dec 1;133(6):1173-1183. doi: 10.1097/ALN.0000000000003550. PMID 32902572
- [Background] Zantek ND, Steiner ME, VanBuren JM, Lewis RJ, Berry NS, Viele K, Krachey E, Dean JM, Nelson S, Spinella PC. Design and logistical considerations for the randomized adaptive non-inferiority storage-duration-ranging CHIlled Platelet Study. Clin Trials. 2023 Feb;20(1):36-46. doi: 10.1177/17407745221126423. Epub 2022 Dec 21. PMID 36541257
- [Derived] Lewis AR, Peffley N, Klompas AM, Ashrani AA. Role of individual factor X concentrate pharmacokinetic studies in perioperative management of AL amyloidosis-associated acquired factor X deficiency. Transfusion. 2023 Sep;63(9):1773-1777. doi: 10.1111/trf.17477. Epub 2023 Jul 10. PMID 37427705
- [Derived] Klompas AM, Stubbs J. Massive transfusion protocol: What's in a name? Transfusion. 2023 Apr;63(4):896-897. doi: 10.1111/trf.17297. No abstract available. PMID 37038736

DOCUMENTS (1):
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT04834414/ICF_001.pdf